CLINICAL TRIAL: NCT03392298
Title: Investigation of Signal Pathway Induced by Colla Corri Asini Regulating Globin Level in Beta Thalassemia Patients With Pregnancy Anemia
Brief Title: Study on the Mechanism of Colla Corri Asini in the Treatment of Thalassemia Patients With Pregnancy Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yanfang Li, associate chief physician, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TH-3
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Thalassemia; Pregnancy
Keywords: Thalassemia; Pregnancy; Globin expression; Colla corii asini
MeSH Terms: conditions — Thalassemia | interventions — colla corii asini

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCA group (Experimental): Participants in CCA group will be treated with 15g of Colla corii asini granule( produced by Dong-E E-Jiao Co., Ltd)， once daily for 4 weeks.
  Interventions: Drug: Colla corii asini
- Control group (No Intervention): Participants in Control group will be treated with nothing, but followed up for 4 weeks.

INTERVENTIONS:
Drug: Colla corii asini — 15g Colla corii asini granule, once daily for 4 weeks
  Other Names: donkey-hide gelatin
  Arms: CCA group

SUMMARY:
This study aims to explore the pathways and targets of regulating globin expression, which might be related to Colla corii asini (CCA, E'jiao) treating anemia in pregnant women with β-thalassemia. Firstly, ten pregnant patients who meet inclusion criteria will be randomly assigned to either the treatment group or control group in a 1: 1 ratio. The patients in the treatment group will be given 15 g of CCA daily for 4 weeks and followed up, while the control group will be treated with nothing and followed up in the same period. The transcriptional test and bioinformatics analysis would be conducted to detect and determine the potential pathways and targets of regulating globin expression before and after the treatment. Secondly, sixty pregnant patients who meet inclusion criteria will be randomly assigned to either the treatment group or control group in a 2: 1 ratio. The treatment group and control group respectively received the same treatment and follow-up regimen as the transcriptional study mentioned above. According to the results of the transcriptional study, the target gene signaling pathway molecules, Hb concentration, and the levels of α-、β-、γ- and δ-globin will be detected and compared.

DETAILED DESCRIPTION:
Thalassemia is a type of hemolytic anemia disease caused by genetic defect of synthesis in one or more globin chains. Among all the single genetic disorders, thalassemia has the highest incidence rate in the world and causes heavy burdens on public health system. In China, the southern provinces suffer from high incidence of thalassemia, which is particularly common in the population of Guangdong, Guangxi and Yunnan provinces. Epidemiological studies showed that in Guangdong alone about 17.83 % of the 14,332 pregnant women across 21 regions examined were diagnosed as carriers of thalassemia.

Recent studies showed that after pregnancy, anemia in β-thalassemia patients tends to turn more serious, the risk of adverse pregnancy outcomes accordingly increase. Currently, no consensus has been reached in treating pregnant thalassemia patients due to lack of safe and effective treatment. Regulation of globin gene expression is the key link of β-thalassemia treatment, but the accessible western medicines have many limitations, including bone marrow suppression, carcinogenicity and teratogenicity, and are not suitable for pregnant patients.

In China, Colla corii asini (CCA, E'jiao) is a gelatin-like traditional Chinese medicine refined from donkey hide and has been widely used in clinical antanemic therapy for more than 2000 years. In the last decade, many studies had addressed the effect of CCA on the anemia using modern pharmacological approaches. The results indicated that CCA contains collagen protein,glycogen and a variety of trace elements, a variety of amino acids, etc. the main components of CCA can promote hematopoiesis by a number of mechanisms which eventually increase the peripheral erythrocyte counts and Hb concentration. Therefore, the investigators proposed that the hematopoietic effects of CCA might also contribute to the treatment of thalassemia with insuffcient or abnormal Hb concentration.

Our previous clinical study showed that CCA can significantly increase the level of hemoglobin and adult hemoglobin (HbA,α2β2) in the pregnant women with β-thalassemia, it was speculated that CCA might induce β globin gene expression, which would be more beneficial to pregnant women than the γ globin gene inducer. But its regulatory pathway is not clear.

This study is designed to explore the pathways and targets of regulating globin expression by using the transcriptomics method, which might be related to CCA treating pregnant anemia in β-thalassemia patients. And then the results of transcriptomics study will be further verified by expanding the clinical samples and implementing cell experiments, aiming to explore the mechanisms of CCA in treating β-thalassemia with pregnant anemia by regulating globin expression.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women diagnosed as minor or intermediate β-thalassemia by genetic tests;
2. Patients with mild anemia (70 g/L≤ Hb<100 g/L) prior to study enrollment;
3. Singleton pregnancy ;
4. Gestational age between 24-32 weeks;
5. Patients having not received blood transfusion in the last 12 weeks;
6. Written informed consent of the patient.

Exclusion Criteria:

1. Known history of allergy or reaction to any component of the investigational product;
2. Allergic to two or more drugs;
3. Patients with severe thalassemia;
4. Anaemia not caused by thalassemia (e.g., iron deficiency, aplastic, megaloblastic or haemolytic anaemia) or bone marrow diseases, leukemia;
5. Twin or multiple pregnancies;
6. Patients having received hemopoietic factors or treated by hematopoietic stem cell transplantation in the last 2 months;
7. Hypersplenism or hypertensive disorder in pregnancy;
8. Patients with any of the following abnormalities: immunodeficiency, primary diseases involving cardiovascular system, liver, kidney, gastrointestinal tract, endocrine system and hematological system;
9. Patients with mental illness;
10. Patients who suffer from drug or alcohol abuse;
11. Patients who addicted to smoking and drinking;
12. Participation in any clinical investigational drug study within the previous 3 months.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin(Hb) | baseline and week 4
  the change of hemoglobin(g/L)

SECONDARY OUTCOMES:
the level of α-、β-、γ- and δ-globin mRNA | baseline and week 4
  the change of α-、β-、γ- and δ-globin mRNA(cycle threshold value)
target gene signaling pathway molecules | baseline and week 4
  the change of gene expression level(fold change)

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Li, PhD, Principal Investigator — the first affiliated hospital of Guangzhou University of Chinese Medicine, Guangzhou
Locations (1):
- the first affiliated hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, He H, Yang L, Li X, Li D, Luo S. Therapeutic effect of Colla corii asini on improving anemia and hemoglobin compositions in pregnant women with thalassemia. Int J Hematol. 2016 Nov;104(5):559-565. doi: 10.1007/s12185-016-2069-0. Epub 2016 Jul 25. PMID 27456464
- [Background] Cheng YL, Zhang XH, Sun YW, Wang WJ, Fang SP, Wu ZK. Clinical Effect and Mechanism of Yisui Shengxue Granules in Thalassemia Patients with Mild, Moderate, or Severe Anemia. Evid Based Complement Alternat Med. 2016;2016:1713897. doi: 10.1155/2016/1713897. Epub 2016 Feb 2. PMID 26949404